CLINICAL TRIAL: NCT01438658
Title: Assessing the Clinical Effectiveness of Serum Biomarkers in the Diagnosis of Metastatic Uveal Melanoma
Acronym: UM
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 001-HMO-CTIL
Record Dates: First submitted 2011-09-15; First posted 2011-09-22 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; metastatic uveal melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sera from patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: A cohort of all the patients.

SUMMARY:
Uveal melanoma is the most common primary intraocular tumor in adults. The local treatment is effective, but patients still die of metastatic disease. It has been shown that early diagnosis of a few isolated metastases can result in a clean surgical excision of the metastases and an extension of the expected survival from 7-12 months to over 10 years on some patients.

Many serum biomarkers are employed in Oncology. It makes sense to try the relevant ones in the diagnosis of metastatic uveal melanoma.

The investigators hypothesis is that a soluble serum biomarker level changes upon development of metastatic disease either by secretion by the tumor cells themselves or by their environment. Detection of changes in biomarker level may lead to the diagnosis of metastases before they can be detected by imaging modalities, thus allowing for early treatment of the metastases and a better chance of success.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of uveal melanoma

Exclusion Criteria:

* refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with uveal melanoma being treated at our center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2011-09; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Significant increase in biomarker level that could be linked with detection of metastases by imaging | up to 12 months before diagnosis of metastases
  Serum will be taken on every clinic visit from the day of diagnosis and on. Change in biomarker level will be assessed from one visit to the previous one, and correlated with imaging information on detection of metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Frenkel, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Specialized Ocular Oncology Service, Hadassah-Hebrew-University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Frenkel S, Nir I, Hendler K, Lotem M, Eid A, Jurim O, Pe'er J. Long-term survival of uveal melanoma patients after surgery for liver metastases. Br J Ophthalmol. 2009 Aug;93(8):1042-6. doi: 10.1136/bjo.2008.153684. Epub 2009 May 7. PMID 19429579
- [Background] Mariani P, Piperno-Neumann S, Servois V, Berry MG, Dorval T, Plancher C, Couturier J, Levy-Gabriel C, Lumbroso-Le Rouic L, Desjardins L, Salmon RJ. Surgical management of liver metastases from uveal melanoma: 16 years' experience at the Institut Curie. Eur J Surg Oncol. 2009 Nov;35(11):1192-7. doi: 10.1016/j.ejso.2009.02.016. Epub 2009 Mar 28. PMID 19329272
- [Background] Haritoglou I, Wolf A, Maier T, Haritoglou C, Hein R, Schaller UC. Osteopontin and 'melanoma inhibitory activity': comparison of two serological tumor markers in metastatic uveal melanoma patients. Ophthalmologica. 2009;223(4):239-43. doi: 10.1159/000206139. Epub 2009 Mar 6. PMID 19270465